CLINICAL TRIAL: NCT02025348
Title: A Randomised, Open-label, 4-way Crossover Study in Healthy Subjects to Explore the Performance of IntelliCap® by Comparing Pharmacokinetic Profiles of a Probe Drug.
Brief Title: Explore the Performance of IntelliCap.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D1840M00044
Record Dates: First submitted 2013-12-20; First posted 2014-01-01 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Plasma Concentration; Pharmacokinetic Profile
MeSH Terms: interventions — Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A metoprolol 50mg (Experimental): IntelliCap® capsule Release profile 1 filled with metoprolol gastroenteral solution 233 mg/mL (dose 50 mg).
  Interventions: Drug: IntelliCap
- Treatment B metoprolol 50mg (Experimental): IntelliCap® capsule Release profile 2 filled with metoprolol gastroenteral solution 233 mg/mL (dose 50 mg).
  Interventions: Drug: IntelliCap
- Treatment C metoprolol 50mg (Experimental): IntelliCap® capsule Release profile 3 filled with metoprolol gastroenteral solution 233 mg/mL (dose 50 mg).
  Interventions: Drug: IntelliCap
- Treatment D metorpolol 50mg (Experimental): metoprolol oral solution 1 mg/mL (dose 50 mg).
  Interventions: Drug: IntelliCap

INTERVENTIONS:
Drug: IntelliCap — Drug release from the IntelliCap® system will be actuated post-gastric emptying of IntelliCap® capsule.
  Other Names: IntelliCap and metoprolol

SUMMARY:
This is an open-label, randomised, 4-way crossover study in twelve healthy male volunteers.

The study will characterise the performance of IntelliCap® by evaluating the plasma concentration and pharmacokinetic profile of a probe drug (IMP; metoprolol) released from IntelliCap® with three different release profiles and the plasma concentration and pharmacokinetic profile of the same probe drug after a single dose of an oral solution.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged between 18 and 50 years of age, inclusive.
* Subjects with a body weight of at least 50 kg and no more than 100 kg, inclusive.
* Subjects with a body mass index (BMI) of 18 - 30 kg/m2, inclusive. BMI = Body weight (kg) / [Height (m)]2.
* Subjects with suitable veins for cannulation or repeated venepuncture.
* Subjects must be available to complete the study.
* Subjects must satisfy a medical examiner about their fitness to participate in the study.
* Subjects must provide written informed consent to participate in the study.

Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* Abnormal vital signs, after 10 min supine rest, defined as any of the following:
* Systolic blood pressure < 100 mmHg or ≥ 140 mmHg.
* Diastolic blood pressure < 50 mmHg or ≥ 90 mmHg.
* Heart rate < 50 or > 85 beats per minute.
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting ECG.
* History of severe allergy/hypersensitivity or on-going clinically important allergy/ hypersensitivity as judged by the Investigator or known hypersensitivity to metoprolol (including other beta-blockers) or any other component of the product.

  •Plasma donation within one month of screening or any blood donation/blood loss greater than 500 mL during the three (3) months prior to screening.
* Receipt of a new chemical entity (defined as a compound which has not been approved for marketing) or participation in any other clinical study that includes drug treatment within at least three (3) months of the first administration of study treatment in this study. The period of exclusion begins three months after the final dose. Note: subjects consented and screened, but not randomised in this study or a previous phase I study, are not excluded.
* Previous randomisation to treatment in the present study.
* Involvement of any CRO/third party contractor or AZ employee and their close relatives regardless of their role.
* Judgement by the Investigator that the subject should not participate in the study if they have any on-going or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.
* Subjects who cannot communicate reliably with the Investigator.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
In vivo performance | Pre-dose, pre-actuation (except in study period when subjects are dosed with oral solution) , 0.5 h, 1 h, 1.5 h, 2 h, 3 h, 4 h, 5 h, 6 h, 7 h, 8 h, 10 h, 12 h, 14 h, 24 h, 28 h, and 32 h
  To assess the in vivo performance of the IntelliCap® system by characterizing the plasma concentration of a probe drug (metoprolol)

SECONDARY OUTCOMES:
Pharmacokinetic parameters | Pre-dose, pre-actuation (except in study period when subjects are dosed with oral solution) , 0.5 h, 1 h, 1.5 h, 2 h, 3 h, 4 h, 5 h, 6 h, 7 h, 8 h, 10 h, 12 h, 14 h, 24 h, 28 h, and 32 h.
  To determine the pharmacokinetic parameters of a probe drug (metoprolol), by assessment of AUC0-t, AUC0-∞, Cmax, tmax, t1/2 and Vz/F.

OTHER OUTCOMES:
Safety | At the end of study, approximately 8 weeks after recruitment.
  Incidence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Febbraro, MD PhD, Principal Investigator — Simbec Research
Locations (1):
- Research Site, Merthyr Tydfil, United Kingdom

REFERENCES:
- See also: D1840M00044_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2726&filename=D1840M00044_CSR_Synopsis.pdf
- See also: Publication — http://www.ncbi.nlm.nih.gov/pubmed/26385166